CLINICAL TRIAL: NCT00219986
Title: A Phase I/II Single Site Open Label Trial of the Safety and Antiviral Activity of C2F5, C2G12, and C4E10 Monoclonal Antibody Infusions in Well-Suppressed HAART-Treated Individuals Treated During Acute and Early HIV-1 Infection
Brief Title: Phase I/II, Open-Label Trial of Three Monoclonal Antibodies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMA 520
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-07-18 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; HIV
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Potent HAART during acute or early HIV-1 infection

SUMMARY:
Monoclonal antibody infusions will prevent rebound of viremia in well-suppressed HAART-treated individuals who began therapy during acute and early HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria: HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. Acute or early HIV-1 infection at the time of HAART initiation defined by HIV-1 RNA detectable with a negative serology or a negative detuned ELISA. HAART for at least 15 months and no more than 1 detectable HIV-1 RNA value (above the 50 copy/mL) for at least 6 months prior to screening.

Laboratory values

* Absolute neutrophil count (ANC) equal to or greter than 750/mm3.
* Hemoglobin equal to or greater than 9.5 g/dL.
* Platelet count equal to or greater than 50,000/mm3.
* Calculated creatinine clearance (CrCl) equal to or greater than 80 mL/min according to the Cockcroft-Gault formula:

Men: (140-age in years) x (wt in kg) = CrCl (mL/min) 72 x (serum creatinine in mg/dL)

Female: (140-age in years) x (wt in kg) x 0.85 = CrCl (mL/min) 72 x (serum creatinine in mg/dL)

* AST (SGOT), ALT (SGPT), and alkaline phosphatase equal to or less than 5 x ULN.
* Total bilirubin equal to or less than 2.5 x ULN.
* Serum Lipase equal to or less than 1.5 x ULN

Negative serum pregnancy test within 14 days. All females of childbearing potential must agree to practice active birth control measures (barrier methods such as condoms, diaphragms, cervical cap, etc. or an intrauterine device such as a coil) to avoid pregnancy while receiving the study drugs and for 30 days after the last dose of the study drugs. Additionally, men enrolled in the study should practice active birth control for the same period of time with their female partners of childbearing potential.

Men and women age >18 years. Ability and willingness of subject to give written informed consent -

Exclusion Criteria:

More than 1 detectable HIV-1 RNA value (>50 copies/mL) within 6 months of screening visit

Pregnancy and breast-feeding.

Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.

Serious illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 30 days prior to study entry.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2003-10; Study Completion 2005-09

PRIMARY OUTCOMES:
To determine the antiviral activity of the combination of 3 monoclonal antibody infusions as an adjunct to HAART

SECONDARY OUTCOMES:
To determine the safety of the combination of 3 monoclonal antibody infusions as an adjunct to HAART

CONTACTS AND LOCATIONS:
Overall Officials: Martin Markowitz, MD, Principal Investigator — Rockefeller University; Saurabh Mehandru, MD, Principal Investigator — Rockefeller University Hosp;ital; Anita Shet, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.rucares.org/clinicalstudies/list.php